CLINICAL TRIAL: NCT03434743
Title: Effect of Non-nutritive Sucking on the Breast to Enhance Breastfeeding in Infants Who Are Born Prematurely
Brief Title: Non-nutritive Sucking and Breastfeeding in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Sandra Fucile (Other)
Responsible Party: Sponsor-Investigator, Dr. Sandra Fucile, Assistant Professor-adjunct, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6021151
Record Dates: First submitted 2018-01-29; First posted 2018-02-15 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Infant,Premature; Infant Development; Infant, Very Low Birth Weight
Keywords: oral feeding; early intervention; premature infant; sucking
MeSH Terms: conditions — Premature Birth | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor, responsible for data collection and follow up interview post hospitalization, is blind to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitative Intervention (Experimental): Experimental rehabilitative intervention consists of non-nutritive sucking on emptied breast, one time per day for 10 minutes.
  Interventions: Other: Rehabilitative
- Control Intervention (Active Comparator): Control active comparator intervention consists of non-nutritive sucking on a pacifier, one time per day for 10 minutes.
  Interventions: Other: Active Comparator

INTERVENTIONS:
Other: Rehabilitative — Non-nutritive sucking on emptied breast
  Arms: Rehabilitative Intervention
Other: Active Comparator — Non-nutritive sucking on pacifier
  Arms: Control Intervention

SUMMARY:
The main objective of this study is to assess whether non-nutritive sucking on an emptied breast will lead to more success with direct breastfeeding than non-nutritive sucking on a pacifier in preterm infants.

DETAILED DESCRIPTION:
Breast milk is vital in the nourishment of premature infants. Early interventions which focus on enhancing infants' oral motor skills required for breastfeeding are needed. There is very limited evidence on early interventions aimed at maintaining rudimentary sucking skills needed for breastfeeding in this high risk population. The main objective of this study is to assess whether non-nutritive sucking on an emptied breast will enhance breast feeding performance in preterm infants.

The target population will consist of clinically stable preterm infants born less born less than or equal to 34 weeks gestational age and whose mother's intention are to breastfeed. Infants will be randomized into the non-nutritive sucking on emptied breast or pacifier group. Both interventions will be administered by mothers. Time to transition to full oral feeding, breastfeeding acquisition at hospital discharge and breastfeeding duration at six months of age will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* born less than or equal to 34 weeks gestational age (GA);
* appropriate size for their GA;
* receiving nasal continuous positive airway pressure;
* receiving only enteral feedings (orogastric or nasogastric);
* mothers are pumping their milk.

Exclusion Criteria:

* congenital anomalies
* mother not expressing milk
* transferred in hospital

Max Age: 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Number of days to transition from full tube to full oral feeds | Through study completion, an average of 2 years
  Number of days to transition from full tube to full oral (bottle/breast) feedings

SECONDARY OUTCOMES:
Breastfeeding acquisition at hospital discharge | Through study completion, an average of 2 years
  Number of infants receive greater than 50% of direct breastfeeding at hospital discharge
Breastfeeding duration | Through study completion, an average of 2 years
  Number of infants receiving direct breastfeeding 6 months after hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fucile S, Wener E, Dow K. Enhancing breastfeeding establishment in preterm infants: A randomized clinical trial of two non-nutritive sucking approaches. Early Hum Dev. 2021 May;156:105347. doi: 10.1016/j.earlhumdev.2021.105347. Epub 2021 Mar 10. PMID 33714801